CLINICAL TRIAL: NCT02257372
Title: A Randomized, Parallel Group Study to Evaluate the Effect of Umeclidinium (UMEC) Added to Inhaled Corticosteroid/ Long-acting Beta-agonist Combination Therapy in Subjects With Chronic Obstructive Pulmonary Disease COPD
Brief Title: A Study to Evaluate the Effect of Umeclidinium (UMEC) as Combination Therapy in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201314
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Results first posted 2015-11-24 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: FEV1; DPI; ICS/LABA; UMEC; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UMEC (62.5 mcg) (Experimental): Participants will self-administer blinded UMEC (62.5 mcg) each morning (once daily) as one inhalation from the double-blind DPI over a treatment period of 12 weeks. Participants will receive open labeled ICS/LABA medication through out duration of the treatment period as background treatment.
  Interventions: Drug: UMEC DPI; Drug: ICS/LABA medication; Drug: Albuterol/salbutamol Metered Dose Inhaler (MDI)
- Placebo (Experimental): Participants will self-administer blinded placebo each morning (once daily) as one inhalation from the double-blind DPI over a treatment period of 12 weeks. Participants will receive open labeled ICS/LABA medication through out duration of the treatment period as background treatment
  Interventions: Drug: Placebo DPI; Drug: ICS/LABA medication; Drug: Albuterol/salbutamol Metered Dose Inhaler (MDI)

INTERVENTIONS:
Drug: UMEC DPI — The UMEC DPI will contain one blister strip which will have 30 blisters of UMEC as dry powder blended with lactose and magnesium stearate, with no companion strip. Each actuation of the DPI will deliver the contents of one blister from each strip simultaneously.
  Arms: UMEC (62.5 mcg)
Drug: Placebo DPI — The matching placebo DPI, identical in appearance to the inhaler containing active study medication, will have two blister strips, each containing 30 blisters of lactose and magnesium stearate.
  Arms: Placebo
Drug: ICS/LABA medication — Participants will use ICS/LABA combinations that are approved for the treatment of COPD at approved doses and frequency including SERETIDE 500/50mcg twice daily, FSC 500/50 mcg twice daily generic products such as AIRFLUSAL FORSPIRO inhaler 500/50mcg twice daily or ROLENIUM ELPENHALER inhaler 500/50mcg twice daily and SYMBICORT TURBUHALER inhaler at doses of 200/6mcg twice daily and 400/12mcg twice daily. The ICS/LABA will be sourced from local commercial stock while on the study
Drug: Albuterol/salbutamol Metered Dose Inhaler (MDI) — Albuterol/salbutamol MDI or nebules will be issued throughout the study as rescue medication, for use as-needed. Albuterol/salbutamol will be sourced from local commercial stock or provided centrally from GlaxoSmithKline.

SUMMARY:
This is a multicenter, randomized, double-blind, parallel-group study to evaluate the efficacy and safety of the addition of UMEC (62.5 microgram[mcg]) when administered once-daily via dry powder inhaler (DPI) to Inhaled corticosteroid/ Long-acting beta2-agonist (ICS/LABA) twice-daily compared with placebo via DPI added to the ICS/LABA therapy over a treatment period of 12 weeks in subjects with COPD. This study is designed to investigate the addition of UMEC to ICS/LABA combinations at approved doses and frequencies for the treatment of COPD including SERETIDE™ 500/50 mcg twice daily, Fluticasone Propionate/Salmeterol Combination (FSC) 500/50 twice daily generic products such as AIRFLUSAL FORSPIRO inhaler 500/50 mcg twice daily or ROLENIUM ELPENHALER inhaler 500/50 mcg twice daily and SYMBICORT TURBUHALER inhaler at doses of 200/6 mcg twice daily and 400/12 mcg twice daily, over 12 weeks in subjects with COPD. Albuterol/salbutamol metered-dose-inhaler (MDI) or nebules will be issued throughout the study for use as-needed (prn).

Subjects who meet the eligibility criteria will be randomly assigned to one of the following blinded study treatment regimens in equal proportion (1:1): UMEC 62.5 mcg once-daily and Placebo once-daily. Approximately 230 subjects (115 subjects per treatment) will be randomized in order to complete at least 206 evaluable subjects. The total duration of the study will be approximately 14 weeks for each subject.

UMEC is a Long-acting Muscarinic Antagonist (LAMA) currently under development as a monotherapy, as a combination product with a LABA, vilanterol (VI), for the treatment of COPD, and as a combination product with an ICS, fluticasone furoate (FF), for the treatment of asthma. The UMEC/VI combination 62.5/25 .mcg once-daily has been approved in the United States (U.S.) and Canada for COPD under the trade name ANORO™ ELLIPTA™ and is under regulatory review in other countries.

SERETIDE, ANORO, and ELLIPTA are trade marks of the GlaxoSmithKline Group of Companies. Other company or product names mentioned herein may be the property of their respective owners.

ELIGIBILITY:
Inclusion Criteria:

* Type of subject: Outpatient.
* Informed Consent: A signed and dated written informed consent prior to study participation.
* Age: Subjects 40 years of age or older at Visit 1.
* Gender: Male and female subjects are eligible to participate in the study. A female is eligible to enter and participate in the study if she is of: Non-child bearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile). Surgically sterile females are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Post-menopausal females are defined as being amenorrhoeic for greater than 1 year with an appropriate clinical profile, e.g., age appropriate, >45 years, in the absence of hormone replacement therapy. OR Child bearing potential, has a negative pregnancy test at screening, and agrees to one of the following acceptable contraceptive methods used consistently and correctly (i.e., in accordance with the approved product label and the instructions of the physician for the duration of the study - screening to follow-up contact): Abstinence; Oral Contraceptive, either combined or progestogen alone; Injectable progestogen; Implants of levonorgestrel; Estrogenic vaginal ring; Percutaneous contraceptive patches; Intrauterine device (IUD) or intrauterine system (IUS) that meets the Standard Operating Procedure (SOP) effectiveness criteria as stated in the product label; Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject. For this definition, "documented" refers to the outcome of the investigator's/designee's medical examination of the subject or review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records; Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository)
* Diagnosis: An established clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society
* Smoking History: Current or former cigarette smokers with a history of cigarette smoking of >=10 pack-years [number of pack years = (number of cigarettes per day / 20) x number of years smoked (e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years)]. Former smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1. Pipe and/or cigar use cannot be used to calculate pack year history.
* Severity of Disease: A pre and post-albuterol/salbutamol Forced Expiratory Volume in One Second /Forced Vital Capacity (FEV1/FVC) ratio of <0.70 and post-albuterol/salbutamol FEV1 of <=70% of predicted normal values at Visit 1 (Screening) calculated using reference values provided by Quanjer.
* Current clinically prescribed medication: The subject must be on the dose and frequency of one of the following ICS/LABA combinations approved for COPD at least 30 days prior screening : FSC at a dose of 500/50 mcg twice-daily (i.e. SERETIDE DISKUS™ inhaler or approved generic product such as AIRFLUSAL FORSPIRO inhaler 500/50 mcg twice daily or ROLENIUM ELPENHALER inhaler 500/50 mcg twice daily) ; The combination of budesonide/formoterol (i.e., SYMBICORT TURBUHALER inhaler) at doses of 200/6 mcg twice-daily or 400/12 mcg twice-daily .
* Dyspnea: A score of >=2 on the Modified Medical Research Council (mMRC) Dyspnea Scale at Visit 1.

Exclusion Criteria:

* Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Asthma: A current diagnosis of asthma.
* Other Respiratory Disorders: Known alpha-1 antitrypsin deficiency, active lung infections (such as tuberculosis), and lung cancer are absolute exclusionary conditions. A subject who, in the opinion of the investigator, has any other significant respiratory conditions in addition to COPD should be excluded. Examples may include clinically significant bronchiectasis, pulmonary hypertension, sarcoidosis, or interstitial lung disease.
* Other Diseases/Abnormalities: The subject is considered unlikely to survive the duration of the study period or has any rapidly progressing disease or immediately life-threatening illness e.g. cancer.
* Contraindications: Any history of allergy or hypersensitivity to any anticholinergic/muscarinic receptor antagonist, beta2-agonist, sympathomimetic, corticosteroid (intranasal, inhaled or systemic) lactose/milk protein or magnesium stearate.
* Hospitalization: Hospitalization for COPD or pneumonia within 12 weeks prior to Visit 1.
* Lower respiratory tract infection: Subjects with lower respiratory tract infection that required the use of antibiotics within 6 weeks prior to Visit 1.
* Lung Resection: Subjects with lung volume reduction surgery within the 12 months prior to Visit 1.
* Unstable or life threatening cardiac disease: UMEC should be used with caution in subjects with severe cardiovascular disease. In the opinion of the investigator, use should only be considered if the benefit is likely to outweigh the risk in conditions such as: Myocardial infarction or unstable angina in the last 6 months; Unstable or life threatening cardiac arrhythmia requiring intervention in the last 3 months; New York Heart Association (NYHA) Class IV heart failure
* 12-Lead Electrocardiogram (ECG): Investigators will be provided with ECG reviews conducted by a centralized independent cardiologist to assist in evaluation of subject eligibility. The Principle Investigator will determine the clinical significance of each abnormal ECG finding in relation to the subject's medical history and exclude subjects who would be at undue risk by participating in the trial. Subjects with the following abnormalities are excluded from participation in the study: Atrial fibrillation with rapid ventricular rate >120 beats per minute (bpm); Sustained or nonsustained ventricular tachycardia; Second degree heart block Mobitz type II and third degree heart block (unless pacemaker or defibrillator had been inserted)
* Antimuscarinic effects: Subjects with medical conditions such as narrow-angle glaucoma, prostatic hypertrophy, or bladder neck obstruction should only be included if, in the opinion of the study physician, the benefit outweighs the risk.
* Interactions: Concomitant administration with beta-blockers and strong Cytochrome P450 3A4 (CYP3A4) inhibitors is only permitted if, in the Investigator's opinion, the likely benefit outweighs the potential risk.
* Severe Hepatic Impairment: Patients with severe hepatic impairment (Child-Pugh class C) should be excluded unless, in the opinion of the investigator, the benefit is likely to outweigh the risk.
* Medication Prior to Spirometry: Unable to withhold albuterol/salbutamol for the 4 hour period required prior to spirometry testing at each study visit.
* Medications Prior to Screening: Use of the following medications according to the following defined time intervals prior to Visit 1: Depot corticosteroids (12 weeks), Systemic, oral or parenteral corticosteroids (6 weeks); Antibiotics (for lower respiratory tract infection) (6 weeks); CYP3A4 strong inhibitors (6 weeks) ; ICS /LABA combination products except SERETIDE and approved FSC 500/50 generic products and SYMBICORT at approved doses and frequencies for COPD (30 days) ; SERETIDE, approved FSC 500/50 generic products, and SYMBICORT at approved doses and frequencies for COPD (12 hours prior to screening); Phosphodiesterase 4 (PDE4) Inhibitor (roflumilast) (14 days); Long-acting muscarinic antagonists (tiotropium, aclidinium, glycopyrronium, UMEC) (7 days); Inhaled long acting beta2 agonists (LABA) (salmeterol, formoterol: 48 hrs) olodaterol, indacaterol (14 days); LAMA/LABA combination products (Apply whichever mono component has the longest washout) Theophyllines (48 hours); Oral beta2-agonists (Long-acting: 48 hours) (Short-acting: 12 hours); Inhaled short acting beta2-agonists (4 hours); Inhaled short-acting anticholinergics (4 hours); Inhaled short-acting anticholinergic/short-acting beta2-agonist combination products (4 hours); Any other investigational medication (30 days or within 5 drug half-lives, whichever is longer). Note: Use of study provided albuterol/salbutamol is permitted during the study, except in the 4-hour period prior to spirometry testing. Intra-articular and epidural corticosteroid injections are permitted. Corticosteroids for short term treatment of COPD exacerbations is allowed
* Oxygen: Use of long-term oxygen therapy (LTOT) described as oxygen therapy prescribed for greater than 12 hours a day. As-needed oxygen use (i.e., <=12 hours per day) is not exclusionary.
* Nebulized Therapy: Regular use (prescribed for use every day, not for as-needed use) of short-acting bronchodilators (e.g., albuterol/salbutamol) via nebulized therapy.
* Pulmonary Rehabilitation Program: Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Visit 1, or who will enter the acute phase of a pulmonary rehabilitation program during the study. Subjects who are in the maintenance phase of a pulmonary rehabilitation program are not excluded.
* Drug or Alcohol Abuse: A known or suspected history of alcohol or drug abuse within 2 years prior to Visit 1.
* Affiliation with Investigator Site: A subject will not be eligible for this study if he/she is an immediate family member of the participating investigator, subinvestigator, study coordinator, or employee of the participating investigator.
* Inability to read: In the opinion of the investigator, any subject who is unable to read and/or would not be able to complete a questionnaire.

DISKUS is a trade mark of the GlaxoSmithKline Group of Companies. Other company or product names mentioned herein may be the property of their respective owners.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2014-09-30 (Actual); Primary Completion 2015-03-24 (Actual); Study Completion 2015-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (25):
- Czechia (5):
  - GSK Investigational Site, Kuřim
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Rokycany
  - GSK Investigational Site, Teplice
  - GSK Investigational Site, Žatec
- Germany (8):
  - GSK Investigational Site, Dillingen an der Donau, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
- Greece (6):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Heraklion, Crete
  - GSK Investigational Site, Kavala
  - GSK Investigational Site, N. Efkarpia, Thessaloniki
  - GSK Investigational Site, Rethymnon, Crete
  - GSK Investigational Site, Thessaloniki
- Netherlands (6):
  - GSK Investigational Site, Almelo
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Harderwijk
  - GSK Investigational Site, Hoorn
  - GSK Investigational Site, Kloosterhaar

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Sousa AR, Riley JH, Church A, Zhu CQ, Punekar YS, Fahy WA. The effect of umeclidinium added to inhaled corticosteroid/long-acting beta2-agonist in patients with symptomatic COPD: a randomised, double-blind, parallel-group study. NPJ Prim Care Respir Med. 2016 Jun 23;26:16031. doi: 10.1038/npjpcrm.2016.31. PMID 27334739
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 201314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 201314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 201314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 201314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 201314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 201314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 201314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants had used one of the following inhaled corticosteroids (ICS)/long-acting beta2-agonist (LABA) combinations for at least 30 days prior to Screening: Fluticasone Propionate/Salmeterol (FSC) 500/50 microgram (mcg) twice-daily (bid); budesonide/formoterol 200/6 mcg bid or 400/12 mcg bid; ICS/LABA combinations per study procedures manual.
Pre-assignment Details: Participants who met eligibility criteria at screening completed an approximately one week run-in period and participants who met the randomisation criteria were entered a 12-week treatment period. A total of 266 participants with chronic obstructive pulmonary disease (COPD) were screened; 236 participants randomized and entered into the study.
Groups:
- Placebo+ICS/LABA: Participants received double-blind placebo via a dry powder inhaler (DPI) once daily and an open-label inhaled corticosteriod (ICS)/Long-acting beta2-agonist(LABA) administered according to the label instructions for 12 weeks. Participants also received albuterol/salbutamol via a metered-dose-inhaler (MDI) or nebules as rescue medication throughout the study for use as needed.
- Umeclidinium 62.5 mcg+ICS/LABA: Participants received Umeclidinium 62.5 microgram(mcg) via a DPI once daily and an open-label ICS/LABA administered according to label instructions for 12 weeks. Participants also received albuterol/salbutamol via a MDI or nebules as rescue medication throughout the study for use as needed.
Period: Overall Study
Arm/Group | Placebo+ICS/LABA | Umeclidinium 62.5 mcg+ICS/LABA
Started | 117 | 119
Completed | 110 | 109
Not Completed | 7 | 10
Not completed — Adverse Event | 3 | 7
Not completed — Lack of Efficacy | 2 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrew consent | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo+ICS/LABA | Umeclidinium 62.5 mcg+ICS/LABA | Total
Number analyzed (Participants) | 117 | 119 | 236
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.1 (7.86) | 65.2 (7.46) | 64.1 (7.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 36 | 78
  Male | 75 | 83 | 158
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Central/South Asian Heritage | 1 | 0 | 1
  White - White/Caucasian/European | 116 | 119 | 235

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in One Second (FEV1) on Day 85
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 on Day 85 is defined as the mean of the FEV1 values obtained 23 and 24 hours after dosing on Day 84 (Week 12). Trough FEV1 was measured using spirometry. BL FEV1 is the mean of the two assessments made 30 and 5 minutes (min) pre-dose on Day 1.Change from BL was calculated as the trough FEV1 value on Day 85 minus the BL value. Analysis was performed using mixed model repeated measures with covariates of treatment, BL FEV1 (mean of the values measured at 30 min and 5 min pre-dose on Day 1), type of ICS/LABA, smoking status, Day, Day by BL interaction and Day by treatment interaction, where Day is nominal.
Time Frame: Baseline (BL) and Day 85
Population: Intent-to-treat (ITT) population: all participants randomized to treatment who received at least one dose of randomized study medication in the treatment period. Only participants with data available at specific timepoint were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo+ICS/LABA | Umeclidinium 62.5 mcg+ICS/LABA
Number analyzed (Participants) | 110 | 109
Liter | -0.033 (0.0184) | 0.090 (0.0183)
Statistical Analysis 1: Comparison: Placebo+ICS/LABA vs Umeclidinium 62.5 mcg+ICS/LABA; Test type: Superiority or Other; p < 0.001, Mixed model repeated measures analysis; Mean Difference (Final Values) = 0.123, 95% CI 2-sided [0.071 to 0.174]

2. Secondary Outcome: Change From Baseline in Weighted Mean 0-6 Hour FEV1 Obtained Post-dose on Day 84
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. The weighted mean FEV1 was derived by calculating the area under the curve, and then dividing the value by the relevant time interval. The weighted mean was calculated by performing six-hour serial spirometry from the pre-dose FEV1 and post-dose FEV1 measurements at 15 minutes, 30 minutes, 1 hour, 3 hours and 6 hours. Baseline FEV1 is the mean of the two assessments made 30 and 5 min pre-dose on Treatment Day 1. Change from Baseline was calculated as weighted mean value on Day 84 minus the Baseline value. Analysis was performed using mixed model repeated measures with covariates of treatment, baseline FEV1 (mean of the values measured at 30 min and 5 min pre-dose on Day 1), type of ICS/LABA , smoking status, Day, Day by baseline interaction and Day by treatment interaction, where Day is nominal.
Time Frame: Baseline and Day 84
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo+ICS/LABA | Umeclidinium 62.5 mcg+ICS/LABA
Number analyzed (Participants) | 110 | 107
Liter | 0.035 (0.0175) | 0.184 (0.0176)
Statistical Analysis 1: Comparison: Placebo+ICS/LABA vs Umeclidinium 62.5 mcg+ICS/LABA; Test type: Superiority or Other; p < 0.001, Mixed model repeated measures analysis; Mean Difference (Final Values) = 0.148, 95% CI 2-sided [0.099 to 0.197]

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study treatment and until the follow up contact (13 weeks).
Description: On-treatment SAEs and non-serious AEs were reported for the ITT Population comprised all subjects randomized to treatment who received at least one dose of randomized study medication in the treatment period.
Arm/Group | Placebo+ICS/LABA | Umeclidinium 62.5 mcg+ICS/LABA
Serious Adverse Events (participants affected / at risk) | 5/117 | 6/119
Other Adverse Events (participants affected / at risk) | 35/117 | 25/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo+ICS/LABA (N=117) | Umeclidinium 62.5 mcg+ICS/LABA (N=119)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Motor neuron disease (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Aortic aneurysm rupture (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo+ICS/LABA (N=117) | Umeclidinium 62.5 mcg+ICS/LABA (N=119)
Nasopharyngitis (Infections and infestations) | 17 | 16
Headache (Nervous system disorders) | 8 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.